CLINICAL TRIAL: NCT04503759
Title: Multicenter Prospective Registry to Evaluate Use and Outcomes of NanoBone in Foot and Ankle Surgery
Brief Title: Artoss Foot and Ankle Surgery Registry
Acronym: ARK
Status: Completed | Type: Observational
Sponsor: Artoss Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HAF002
Record Dates: First submitted 2020-07-30; First posted 2020-08-07 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Arthritis Foot; Trauma Injury; Deformity; Bone
MeSH Terms: conditions — Accidental Injuries; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Foot and Ankle Surgery using NanoBone: All patients in the study will be drawn from the individual surgeons' practice. Patients will be among those already scheduled for foot and ankle surgery after having failed conservative treatment, or will have had foot and ankle surgery using NanoBone products but have not completed their standard of care follow-up as determined by the surgeon's practice. In addition, the surgeon has determined that the use of a NanoBone product is or was clinically necessary for the patient. The choice of a NanoBone product, as well as the surgery, is or was independent of this research project. Only patients who have had NanoBone implanted and consent to participate and meet the inclusion-exclusion criteria will be included in the registry.
  Interventions: Other: NanoBone Bone Graft Substitute

INTERVENTIONS:
Other: NanoBone Bone Graft Substitute — Synthetic, biodegradable bone grafting material that is composed of non-sintered nanocrystalline hydroxyapatite (HA) which is embedded in a silica gel matrix (amorphous SiO2). The ratio of HA/SiO2 has been chosen to optimize the rate of biodegradation for treatment of osseous defects in human bone. NanoBone does not contain any components of animal or human origin, eliminating the possibility of transmission of infection or disease.
  Other Names: nanoHA-SiO2

SUMMARY:
This prospective registry was designed as an observational study to ascertain how commercially available NanoBone products are being used by surgeons performing foot and ankle surgery which involves bone grafting, as well as determining relevant patient outcomes.

DETAILED DESCRIPTION:
This multicenter prospective patient registry was developed with the aim of documenting how surgeons are utilizing NanoBone products in foot and ankle surgery along with relevant patient outcomes. These outcomes include radiographic measures such as fusion or graft consolidation success, instrumentation integrity, and clinical outcomes (symptom and function improvement) based on investigator and patient-based outcome assessments.

The primary objective of this study is to document and analyze the use of NanoBone products in foot and ankle surgery (as a stand-alone bone graft, no other local bone, autograft, bone graft substitute, or biologic product used) and determine both radiographic success and clinical outcomes. All product related adverse events will be documented, tabulated, and summarized.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older.
* Patient is or was diagnosed with a pathology of the foot or ankle, having failed conservative treatment, and surgeon has determined that surgery with bone graft is medically necessary.
* The surgeon has determined that NanoBone is or was clinically indicated.
* NanoBone will be or was used as a stand-alone bone graft (no autograft, other bone graft substitute, or biologic planned or used).
* Patient capable of understanding the content of the Informed Consent Form
* Patient willing and able to participate in the registry protocol including the surgeon's standard follow-up visits and clinical evaluations.
* Patient who has agreed to participate in the registry by providing consent according to the applicable local law and the declaration of Helsinki.

Exclusion Criteria:

* Severe vascular or neurological disease
* Uncontrolled diabetes
* Severe degenerative disease (other than degenerative disc disease)
* Severely impaired renal function
* Hypercalcemia, abnormal calcium metabolism
* Existing acute or chronic infections, especially at the site of the operation
* Inflammatory bone disease such as osteomyelitis
* Malignant tumors
* Patients who are or plan to become pregnant.
* Uncooperative patients who cannot or will not follow post-operative instruction, including individuals who abuse drugs and/or alcohol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the study will be drawn from the individual surgeons' practice. Patients will be among those already scheduled for foot and ankle surgery after having failed conservative treatment, or will have had foot and ankle surgery using NanoBone products but have not completed their standard of care follow-up as determined by the surgeon's practice. In addition, the surgeon has determined that the use of a NanoBone product is or was clinically necessary for the patient. The choice of a NanoBone product, as well as the surgery, is or was independent of this research project. Only patients who have had NanoBone implanted and consent to participate and meet the inclusion-exclusion criteria will be included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Radiographic Success | 6-months
  Fusion/Graft Consolidation: Evidence of bony (osseous) bridging between the graft material and the patient's bone in the segment requiring fusion or reconstruction.

SECONDARY OUTCOMES:
Safety Evaluation | 6-months
  Occurrence of Complications or Adverse Events

OTHER OUTCOMES:
Clinical Success | 6-months
  Change from baseline in Visual Analog Scale (VAS) pain score (0=no pain, 10=worst possible pain
Function | 6-months
  Change from baseline in Foot and Ankle Ability Measure (FAAM)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Cassidy, PhD, Study Director — Artoss Inc.
Locations (8):
- United States (8):
  - Phoenix Foot and Ankle Institute, Scottsdale, Arizona
  - Florida Orthopedic Foot & Ankle Center, Sarasota, Florida
  - Illinois Orthopedic Institute, Joliet, Illinois
  - Morrison Hospital, Morrison, Illinois
  - Podiatry Associates of Indiana, Indianapolis, Indiana
  - Hoosier Foot and Ankle, Kokomo, Indiana
  - The Iowa Clinic, West Des Moines, Iowa
  - Orthopedic Associates of Duluth, Duluth, Minnesota